CLINICAL TRIAL: NCT05975463
Title: Prospective Single Arm, Single Center, Phase II Clinical Study of Hepatic Artery Infusion of Adebrelimab Combined With Bevacizumab Treatment System for Advanced Hepatocellular Carcinoma With Failure of Systemic Therapy Combined With Interventional Therapy
Brief Title: Hepatic Artery Infusion of Adebrelimab Combined With Bevacizumab in the Treatment of Advanced Hepatocellular Carcinoma With Failure of Systemic Therapy Combined With Interventional Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HuiKai Li (Other)
Responsible Party: Sponsor-Investigator, HuiKai Li, Director, Tianjin Medical University Cancer Institute and Hospital
Organization: Tianjin Medical University Cancer Institute and Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1316-HCC-TJ-001
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+Adebrelimab+Bevacizumab (Experimental): hepatic artery infusion of Adebrelimab 1200mg, d1, q3w, combined with hepatic artery infusion of Bevacizumab 5mg/kg, d1, q3w, HAIC treatment for 3-4 times.
  Interventions: Procedure: HAIC; Drug: Adebrelimab; Drug: Bevacizumab

INTERVENTIONS:
Procedure: HAIC — hepatic artery infusion for 3-4 times.
Drug: Adebrelimab — hepatic artery infusion of Adebrelimab 1200mg, d1, q3w，for 3-4 times.
Drug: Bevacizumab — hepatic artery infusion of Bevacizumab 5mg/kg, d1, q3w, for 3-4 times.

SUMMARY:
The goal of this prospective single arm, Phase II Clinical Study is to explore and evaluate the efficacy and safety of hepatic artery infusion of Adebrelimab combined with Bevacizumab in the treatment of patients with advanced hepatocellular carcinoma who failed in systematic therapy combined with interventional therapy.

Participants will receive hepatic artery infusion of Adebrelimab 1200mg, d1, q3w, combined with hepatic artery infusion of Bevacizumab 5mg/kg, d1, q3w, HAIC treatment for 3-4 times.

ELIGIBILITY:
Inclusion Criteria:

* 1. Non resectable advanced hepatocellular carcinoma confirmed by pathological and clinical imaging examinations.
* 2. Patients who have previously received systematic treatment combined with failed or intolerable interventional therapy.
* 3. Male or female, aged ≥ 18 years at the time of signing the Informed consent form (ICF).
* 4. The liver should have at least one measurable target lesion (RECIST v1.1). If it is an active lesion after local treatment (radiotherapy, ablation, transcatheter arterial chemoembolization, etc.), local treatment should be completed 4 weeks before the screening period imaging examination.
* 5. The patient's Eastern Oncology Collaborative Group (ECOG) physical condition score is 0 or 1.
* 6. The patient's organ and blood system functions meet the requirements:

  1. Hematology function: Absolute neutrophil count (ANC) ≥ 1.5 x 10 ^ 9/L, platelet count ≥ 75 x 10 ^ 9/L
  2. Adequate renal function: serum creatinine<1.5x ULN or creatinine clearance rate>40 mL/min (Cockcroft Fault formula)
  3. Liver function: Total bilirubin ≤ 1.5 x ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 5 x ULN
  4. Coagulation function: Within the normal range of Prothrombin time (PT) .
* 7. Female participants with Fertility need to carry out serum pregnancy test within 72 hours before starting the study drug administration, and the result is negative, and take effective contraceptive measures (such as Intrauterine device, contraceptive pill or pregnancy avoidance condom) during the test period and at least 3 months after the last administration; For male participants whose partners are Fertility women, they should be surgically sterilized or agree to take effective contraceptive measures during the trial period and within 3 months after the last administration.
* 8. The participants have good compliance and cooperate with follow-up.

Exclusion Criteria:

* 1. Has a history of allergies to any component of the study drug in the past;
* 2. Known to be allergic to Programmed Death-1/Programmed Death-L1 (PD-1/PD-L1) antibodies or have experienced drug-related Immune related adverse events (irAEs) in the past, in accordance with the "Guidelines Of Chinese Society Of Clinical Oncology [CSCO]Management Of Immune Checkpointinhibitor-Related Toxicity 2019", it meets the indication for permanent discontinuation of medication;
* 3. There are known Contraindication of percutaneous hepatic artery infusion;
* 4. Has received or is currently receiving any of the following treatments in the past:

  1. The patient underwent major surgical procedures within 14 days prior to entering the study (puncture biopsy is not included)
  2. Previous or planned immune therapy such as Chimeric antigen receptor T cell immunotherapy (CAR-T) and vaccines
* 5. Have any active autoimmune disease or history of autoimmune disease, including but not limited to interstitial pneumonia, enteritis, hepatitis, hypophysitis, Vasculitis, nephritis, hyperthyroidism, hypothyroidism (it can be considered to be included after hormone replacement treatment); Patients with psoriasis or childhood asthma/allergy that has completely alleviated and does not need any intervention after adulthood can be considered for inclusion, but patients who need medical intervention with Bronchiectasis cannot be included;
* 6. Poor nutritional status, BMI<18.5 Kg/m2; If symptomatic nutritional support is provided and corrected before enrollment, and evaluated by the main investigator, enrollment can continue to be considered;
* 7. Have a history of immune deficiency, including positive Diagnosis of HIV/AIDS, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation or allogeneic bone marrow transplantation;
* 8. There are clinical symptoms or diseases of the heart that cannot be well controlled, including but not limited to: (1) New York Heart Association (NYHA)grade II or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias that have not undergone clinical intervention or are still poorly controlled after clinical intervention;
* 9. Serious infection (CTCAE>grade 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, Bloodstream infections, infection complications, etc. requiring hospitalization; Baseline chest imaging examination indicates the presence of active pulmonary inflammation, symptoms and signs of infection within 14 days prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, excluding prophylactic use of antibiotics;
* 10. Those who have been found to have active pulmonary tuberculosis infection through medical history or CT examination, or have a history of active pulmonary tuberculosis infection within 1 year before enrollment, or have a history of active pulmonary tuberculosis infection more than 1 year before but have not received formal treatment;
* 11. There is active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL) and hepatitis C (hepatitis C antibody is positive, and HCV RNA is higher than the detection limit of the analytical method);
* 12. Other malignant tumors were diagnosed within 5 years before the first use of the study drug, except for malignant tumors with low risk of metastasis or death (5-year survival rate>90%), such as fully treated skin Basal-cell carcinoma or squamous cell skin cancer or cervical Carcinoma in situ, which can be considered to be included in the group;
* 13. Pregnant or lactating women;
* 14. Previous history of hypertensive crisis or hypertensive encephalopathy;
* 15. Use Nonsteroidal anti-inflammatory drug (NSAIDs) for long-term daily treatment;
* 16. Untreated or incompletely treated esophageal and/or gastric varices with high risk of bleeding or bleeding;
* 17. Previous bleeding events caused by esophageal and/or gastric varices within 6 months prior to the start of the study treatment;
* 18. According to the judgment of the investigators, there are other factors that may lead to forced termination of the study, such as suffering from other serious illnesses (including mental illness) requiring concurrent treatment, alcoholism, drug abuse, family or social factors, which may affect the safety or compliance of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to one year
  Objective response rate

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to two years
  Progression-free survival：The time from the start of treatment to the progression of the disease or death from any cause
Overall Survival (OS) | Up to two years
  Overall Survival：The survival time from enrollment to death from any cause.
Disease Control Rate (DCR) | Up to one year
  Disease Control Rate: Ratio of complete response (CR)+partial response (PR)+stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No